CLINICAL TRIAL: NCT02212106
Title: A Phase IV, Multicenter, Randomized, Observer-blind, Parallel-arm Study to Evaluate the Safety and Tolerability of CSL's Trivalent Influenza Virus Vaccine (CSL TIV) in Children 5 to Less Than 9 Years of Age.
Brief Title: A Study to Evaluate the Safety and Tolerability of Trivalent Influenza Virus Vaccine in Children Aged 5 Years to < 9 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CSLCT-USF-10-69; 2015-000175-27 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) (Experimental): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total haemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  Interventions: Biological: bioCSL Trivalent Influenza Virus Vaccine (CSL TIV)
- Comparator Quadrivalent Influenza Virus Vaccine (Active Comparator): The comparator vaccine is a US-licensed product containing four recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season.
  Interventions: Biological: Comparator Quadrivalent Influenza Virus Vaccine

INTERVENTIONS:
Biological: bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) — Subjects will receive one or two study vaccinations depending on their influenza vaccine history. The vaccine will be administered by intramuscular injection.
  Arms: bioCSL Trivalent Influenza Virus Vaccine (CSL TIV)
Biological: Comparator Quadrivalent Influenza Virus Vaccine — Subjects will receive one or two study vaccinations depending on their influenza vaccine history. The vaccine will be administered by intramuscular injection.
  Other Names: Fluzone Quadrivalent
  Arms: Comparator Quadrivalent Influenza Virus Vaccine

SUMMARY:
This is a study to assess the safety of a bioCSL split virion, inactivated Trivalent Influenza Virus vaccine containing the 2014/2015 Northern Hemisphere strains of vaccine in children aged 5 years to less than 9 years. Comparison will be made to a licensed Quadrivalent Influenza Virus vaccine that complies with the FDA recommendations for the 2014/2015 influenza season in the US.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 5 to less than 9 years at the time of first study vaccination.
* The subject's parent or guardian to provide written informed consent and be willing and able to adhere to all protocol requirements.
* In good health, as determined by medical history and a targeted physical examination (if warranted).

Exclusion Criteria:

* Known hypersensitivity to a previous dose of Influenza Virus Vaccine or allergy to eggs or any components of the study vaccines.
* Clinical signs of significant active infection or an elevated oral temperature at study entry.
* A clinically significant medical or psychiatric condition.
* A history of seizures or febrile convulsions or Guillain-Barré syndrome.
* Vaccination with a seasonal or experimental influenza virus vaccine in the 6 months preceding study entry.
* Vaccination with a licensed vaccine within 14 days preceding study entry, or planning to be vaccinated with another licensed vaccine before the study exit evaluation.
* Currently receiving systemic glucocorticoid therapy (excluding intra-articular, topical or inhaled preparations) or have received such therapy within the 3 months preceding study entry.
* Currently receiving immunoglobulins and/or any blood products or have received such treatment within the 3 months preceding the administration of the study vaccine.
* Currently receiving treatment with warfarin or other anticoagulants.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 402 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: bioCSL Pty Ltd Clinical Program Director, Study Director — Seqirus
Locations (11):
- United States (11):
  - Site 286, Los Angeles, California
  - Site 289, Boise, Idaho
  - Site 287, St Louis, Missouri
  - Site 285, Binghamton, New York
  - Site 290, Durham, North Carolina
  - Site 281, Raleigh, North Carolina
  - Site 280, Winston-Salem, North Carolina
  - Site 284, Charleston, South Carolina
  - Site 283, Austin, Texas
  - Site 282, Fort Worth, Texas
  - Site 288, San Angelo, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 22-SEP-2014, Last Patient In: 15-OCT-2014, Last Patient Last Visit: 05-DEC-2014. Number of activated sites that enrolled subjects: 11 (all based in USA).
Pre-assignment Details: Number of subjects screened: 407 Number of screen failures: 5 (Reason: all due to not meeting inclusion/exclusion criteria).
Groups:
- bioCSL Trivalent Influenza Virus Vaccine (CSL TIV): The bioCSL study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2014/2015 influenza season).
  bioCSL Trivalent Influenza Virus Vaccine (CSL TIV): Subjects will receive one or two study vaccinations depending on their influenza vaccine history. The vaccine will be administered by intramuscular injection.
Period: Overall Study
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Started | 302 | 100
Completed | 292 | 96
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine | Total
Number analyzed (Participants) | 302 | 100 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (1.05) | 6.6 (1.02) | 6.6 (1.04)
Age, Customized [Number; unit: participants]
  Age 5 to < 9 years | 302 | 100 | 402
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 46 | 193
  Male | 155 | 54 | 209
Region of Enrollment [Number; unit: participants]
  United States | 302 | 100 | 402

OUTCOME MEASURES:

1. Primary Outcome: The Frequency and Intensity of Fever Events Occurring During the 7 Days After Each Administration of CSL TIV Vaccine.
Description: The overall percentage of subjects reporting at least one fever event after administration of bioCSL TIV. A fever event was defined as an oral temperature ≥ 38°C (≥ 100.4°F). The intensity was calculated as follows: • Mild: ≥ 100.4 to < 101.3°F (≥ 38.0 to < 38.5°C) • Moderate: ≥ 101.3 to < 102.2°F (≥ 38.5 to < 39.0°C) • Severe: ≥ 102.2°F (≥ 39.0°C)
Time Frame: 7 days after each administration of vaccine.
Population: All randomized subjects who received at least one scheduled vaccination and had post-vaccination follow-up safety data available.
Measure: Number; unit: Percentage of subjects
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV)
Number analyzed (Participants) | 292
Percentage of subjects
  Total | 8.2
  Mild | 4.1
  Moderate | 2.1
  Severe | 2.1

2. Secondary Outcome: The Frequency and Intensity of Fever Events Occurring During the 7 Days After Each Administration of the Comparator Influenza Virus Vaccine.
Description: The overall percentage of subjects reporting at least one fever event after administration of the comparator influenza virus vaccine. A fever event was defined as an oral temperature ≥ 38°C (≥ 100.4°F). The intensity was calculated as follows: • Mild: ≥ 100.4 to < 101.3°F (≥ 38.0 to < 38.5°C) • Moderate: ≥ 101.3 to < 102.2°F (≥ 38.5 to < 39.0°C) • Severe: ≥ 102.2°F (≥ 39.0°C).
Time Frame: 7 days after each administration of vaccine.
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Comparator Quadrivalent Influenza Virus Vaccine
Number analyzed (Participants) | 98
Percentage of subjects
  Total | 9.2
  Mild | 1.0
  Moderate | 4.1
  Severe | 4.1

3. Secondary Outcome: The Frequency and Intensity of Vaccine-related Fever Events Occurring During the 7 Days After Each Administration of CSL TIV Vaccine or Comparator Influenza Virus Vaccine.
Description: Percentage of subjects with a related fever event (overall) by study vaccine group based on the number of subjects contributing any follow up safety information for at least one data value of an individual sign/symptom. Excludes subjects with missing intensity information for the whole 7 days. Mild fever: ≥ 100.4 to < 101.3º F (≥ 38.0 to < 38.5º C). Moderate fever: ≥ 101.3 to < 102.2º F (≥ 38.5 to < 39.0º C). Severe fever: ≥ 102.2º F (≥ 39.0º C).
Time Frame: 7 days after each administration of vaccine.
Population: All randomized subjects who received at least one scheduled vaccination and had post-vaccination followup safety data available.
Measure: Number; unit: Percentage of subjects
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Number analyzed (Participants) | 292 | 98
Percentage of subjects
  Total | 7.5 | 5.1
  Mild | 4.1 | 1.0
  Moderate | 1.7 | 4.1
  Severe | 1.7 | 0

4. Secondary Outcome: The Frequency and Intensity of Solicited Local Adverse Events (AEs) Occurring During the 7 Days After Each Administration of CSL TIV or the Comparator Influenza Virus Vaccine.
Description: The overall frequency and intensity of solicited local Adverse Events (AEs) occurring during the 7 days after each administration of bioCSL TIV or the comparator influenza virus vaccine. Percentage of subjects who experienced each event are based on the number of subjects in the Safety Population group. Excludes subjects with missing intensity information for the whole 7 days. Percentages for intensity are based on the number of subjects with non-missing intensity data. Only the maximum intensity experienced between Day 1 and Day 7 are presented for each subject.
Time Frame: 7 days after each administration of vaccine.
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Number analyzed (Participants) | 292 | 98
Percentage of subjects
  Total | 70.2 | 68.4
  Total - mild | 49.8 | 46.9
  Total - moderate | 17.2 | 15.3
  Total - severe | 3.4 | 6.1
  Pain - total | 64.4 | 57.1
  Pain - mild | 53.3 | 42.9
  Pain - moderate | 9.6 | 13.3
  Pain - severe | 1.7 | 1.0
  Redness - total | 34.9 | 37.8
  Redness - mild | 26.8 | 30.6
  Redness - moderate | 7.2 | 3.1
  Redness - severe | 1.0 | 4.1
  Swelling/Lump - total | 29.8 | 40.8
  Swelling/Lump - mild | 21.0 | 28.6
  Swelling/Lump - moderate | 7.9 | 8.2
  Swelling/Lump - severe | 1.0 | 4.1

5. Secondary Outcome: The Frequency and Intensity of Solicited Systemic AEs Occurring During the 7 Days After Each Administration of CSL TIV or the Comparator Influenza Virus Vaccine.
Description: The overall frequency and intensity of solicited systemic Adverse Events (AEs) occurring during the 7 days after each administration of CSL TIV or the comparator influenza virus vaccine. Percentage of subjects who experienced each event are based on the number of subjects in the Safety Population group. Excludes subjects with missing intensity information for the whole 7 days. Percentages for intensity are based on the number of subjects with non-missing intensity data. Only the maximum intensity experienced between Day 1 and Day 7 are presented for each subject.
Time Frame: 7 days after each administration of vaccine.
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Number analyzed (Participants) | 292 | 98
Percentage of subjects
  Total | 40.8 | 44.9
  Total - mild | 28.4 | 21.4
  Total - moderate | 8.6 | 19.4
  Total - severe | 3.8 | 4.1
  Headache - total | 14.7 | 23.5
  Headache - mild | 11.4 | 12.2
  Headache - moderate | 3.1 | 10.2
  Headache - severe | 0.3 | 1.0
  Malaise - total | 8.9 | 14.3
  Malaise - mild | 7.2 | 9.2
  Malaise - moderate | 1.0 | 5.1
  Malaise - severe | 0.7 | 0
  Muscle ache (myalgia) - total | 24.3 | 23.5
  Muscle ache (myalgia) - mild | 20.0 | 15.3
  Muscle ache (myalgia) - moderate | 3.4 | 7.1
  Muscle ache (myalgia) - severe | 1.0 | 1.0
  Diarrhea - total | 5.1 | 11.2
  Diarrhea - mild | 3.8 | 6.1
  Diarrhea - moderate | 1.0 | 4.1
  Diarrhea - severe | 0.3 | 1.0
  Nausea - total | 6.8 | 9.2
  Nausea - mild | 5.5 | 6.1
  Nausea - moderate | 0.7 | 2.0
  Nausea - severe | 0.7 | 1.0
  Vomiting - total | 2.7 | 2.0
  Vomiting - mild | 2.1 | 0
  Vomiting - moderate | 0.3 | 1.0
  Vomiting - severe | 0.3 | 1.0
  Fever - total | 8.2 | 9.2
  Fever - mild | 4.1 | 1.0
  Fever - moderate | 2.1 | 4.1
  Fever - severe | 2.1 | 4.1

6. Secondary Outcome: The Frequency and Intensity of Unsolicited AEs Occurring During the 7 Days After Each Administration of CSL TIV or the Comparator Influenza Virus Vaccine.
Description: The overall frequency and intensity of unsolicited Adverse Events (AEs) occurring during the 7 days after each administration of CSL TIV or the comparator influenza virus vaccine. Percentage of subjects who experienced each event are based on the number of subjects in the Safety Population group. Excludes subjects with missing intensity information for the whole 7 days. If a subject has multiple events of the same intensity or causality, then they are counted only once in that intensity or causality. However, subjects can be counted more than once overall.
Time Frame: 7 days after each administration of vaccine.
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Number analyzed (Participants) | 292 | 98
Percentage of subjects
  Total | 14.0 | 22.4
  Total - mild | 8.2 | 12.2
  Total - moderate | 5.8 | 10.2
  Total - severe | 0.7 | 1.0

7. Secondary Outcome: The Incidence of Serious Adverse Events (SAEs) Occurring up to 7 Days After the Last Administration of CSL TIV or the Comparator Influenza Virus Vaccine.
Description: The number of subjects experiencing at least one SAE.
Time Frame: 7 days after each administration of vaccine.
Population: as for outcome 3
Measure: Number; unit: Number of subjects
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Number analyzed (Participants) | 292 | 98
Number of subjects | 1 | 0

ADVERSE EVENTS:
Time Frame: 7 days after each vaccination.
Description: Overall data (following first & second vaccination) for Safety Population is shown. If a subject has multiple events of the same intensity or causality, then they are counted only once in that intensity or causality. However, subjects can be counted more than once overall
Arm/Group | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) | Comparator Quadrivalent Influenza Virus Vaccine
Serious Adverse Events (participants affected / at risk) | 1/292 | 0/98
Other Adverse Events (participants affected / at risk) | 222/292 | 75/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) (N=292) | Comparator Quadrivalent Influenza Virus Vaccine (N=98)
Delirium febrile (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | bioCSL Trivalent Influenza Virus Vaccine (CSL TIV) (N=292) | Comparator Quadrivalent Influenza Virus Vaccine (N=98)
Headache (Nervous system disorders) | 43 (55) | 23 (32)
Pain (General disorders) | 188 (230) | 56 (71)
Redness (General disorders) | 102 (117) | 37 (44)
Swelling / lump (General disorders) | 87 (101) | 40 (50)
Malaise (General disorders) | 26 (32) | 14 (18)
Fever (General disorders) | 24 (25) | 9 (11)
Diarrhea (Gastrointestinal disorders) | 15 (19) | 11 (16)
Nausea (Gastrointestinal disorders) | 20 (22) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 71 (80) | 23 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.